CLINICAL TRIAL: NCT05555992
Title: Electrical Activation Mapping Guided Tailor Made Approach for Cardiac Resynchronization Therapy for Non-responder
Brief Title: CardioInsight 2 - Non-responder
Acronym: CardioInsight2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Bryan Ping Yen YAN, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018.215
Record Dates: First submitted 2022-09-15; First posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Device: Electrical Activation Mapping Guided Cardiac resynchronization therapy

INTERVENTIONS:
Device: Electrical Activation Mapping Guided Cardiac resynchronization therapy — To study the feasibility to optimize configuration of CRT delivery for acute correction of electrical dyssynchrony using a noninvasive mapping of global electrical activation

SUMMARY:
Background Cardiac Resynchronization Therapy (CRT) is proven to improve survival and heart function of patient with certain electrical conduction abnormality and heart failure. However, in patient with certain electrical conduction abnormality, being nonresponder is observed in up to 40% in patient receiving CRT. Conventionally the surgical approach of CRT is to implant one pacing lead in the right heart and one in the left heart to resynchronize the contraction and the pacing lead in the left heart is usually placed in the posterior or lateral portion of the left heart. However, this single approach may not be optimal, especially for those patients with conduction abnormality known to have no response to CRT. Purpose of the clinical investigation. The purpose of the Electrical Activation Guided CRT for Nonresponders Study is to study the effectiveness of an addition of Hisbundle pacing approach to CRT nonresponder by direct His-bundle pacing to improve the responder rate of nonresponder of conventional CRT and a tailored made approach to CRT procedure by using a noninvasive globally mapping system studying the electrical conduction under different approaches to delivery CRT. The pacing approach that optimally corrects conduction abnormality will be determined before the actual addition of new lead procedure.

Conduct of the Investigation This study will include 18 patients already implanted with device delivering conventional CRT that known to have no response to the conventional CRT after 6 months of the CRT therapy from Prince of Wales Hospital, Hong Kong. You will be followed in the device clinic as per usual care after your participation in the study is completed.

ELIGIBILITY:
Inclusion Criteria:

* Adult (aged 18 or above) of both sexes
* Ischemic or non-ischemic cause of heart failure
* QRS duration > 120 ms, non -LBBB type of conduction disturbance
* NYHA class III or above
* Informed consent by the patient
* Already received stable dose of guideline directed medical therapy for at least 3 months

Exclusion Criteria:

* LBBB patients
* Pregnant women
* Participation in another study
* Patient with contraindication to left ventricle catheterization by a retrograde aortic approach

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Left Ventricle end systolic volume reduction | 6 months
  The responder rate of greater than 10% of LV end systolic volume reduction measured by echocardiogram.

SECONDARY OUTCOMES:
Electrical desynchrony index | During procedure
  The acute electrical desynchrony indices (the standard deviation of activation times throughout the epicardium) of different methods of CRT delivery. Lower indicate larger improvement.
Hemodynamic response monitoring | During procedure
  Monitor the difference in hemodynamic responses of different methods of CRT delivery. The hemodynamic response will be maximal dp/dt as measured by pressure wire introduced into the left ventricle during the procedure.
Procedure duration of different methods of CRT delivery | During procedure
  Procedure duration of the optimal CRT delivery method as determined by the best improvement in electrical desynchrony indices.
Implantation success rate of different methods of CRT delivery | During procedure
  Implantation success rate of the optimal CRT delivery method as determined by the best improvement in electrical desynchrony indices.
Cine images and chest X ray | 6 months
  Cine images (PA, LAO 300, RAO 300) and Chest X ray (PA view) of patients will be obtained for evaluation of changes in disease
Echocardiogram parameters: left ventricular systolic and diastolic volume | 6 months
  Echocardiogram parameters: left ventricular systolic and diastolic volume at baseline, 3 months and 6 months.
Echocardiogram parameters: left ventricular ejection fraction | 6 months
  Echocardiogram parameters: left ventricular ejection fraction at baseline, 3 months and 6 months
Echocardiogram parameters: degree of mitral regurgitation | 6 months
  Echocardiogram parameter: degree of mitral regurgitation at baseline, 3 months and 6 months.
Echocardiogram parameters: strain imaging | 6 months
  Echocardiogram parameters: strain imaging at baseline, 3 months and 6 months
Change in New York Heart Association (NYHA) class | 6 months
  Overall changes in QoL measured by change in NYHA class at baseline, 3 months and 6 months.
Device set-up parameter: defibrillation threshold | 6 months
  Device parameters including defibrillation threshold at implant and 6 months follow-up.
Post-operation Complication rate | 6 months
  Peri-operative and 6 months follow-up complications rate:
  1. Thromboembolic event
  2. Dislodgement and migration of pacing leads
  3. Phrenic nerve stimulation
  4. Others
Change in 6 minute hall walk test | 6 months
  Compare result of 6 minute hall walk test at baseline, 3 months and 6 months.
Change in HF Patient Global Assessment Questionnaire | 6 months
  Compare result of HF Patient Global Assessment Questionnaire at baseline, 3 months and 6 months.
Change in quality of life | 6 months
  Change in quality of life assessed by Minnesota's living with heart failure (MLWHF) questionnaire at baseline, 3 months and 6 months.
Device set-up parameter: defibrillation sensitivity | 6 months
  Device parameters including defibrillation sensitivity at implant and 6 months follow-up.
Device set-up parameter: lead impedance | 6 months
  Device parameters including lead impedance of pacing leads at implant and 6 months follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Byran Yan, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong